CLINICAL TRIAL: NCT02261337
Title: Do Gait Speed and Markers of Sarcopenia Predict Prognosis in Patients With Chronic Respiratory Disease?
Brief Title: Is Gait Speed and Sarcopenia Prognostic in Chronic Respiratory Disease?
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013LF003H
Record Dates: First submitted 2014-05-01; First posted 2014-10-10 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease and Allied Conditions
Keywords: Sarcopenia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study aims to assess usual walking speed (4-metre gait speed) and markers of sarcopenia predict mortality in patients with chronic respiratory disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic respiratory disease who are able to complete the assessments.

Exclusion Criteria:

* Significant co-morbidities that would limit walking ability, exercise capacity or make exercise unsafe (e.g. unstable ischaemic heart disease, neuromuscular disease, severe hip/lower limb joint pain, peripheral vascular disease, lower limb amputation).
* Any patient whom the Chief Investigator feels it is unsafe to exercise (e.g. unstable cardiovascular disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with chronic respiratory disease. The cohort will be recruited from Harefield hospital.
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Number of participant deaths | 1 year

SECONDARY OUTCOMES:
Number of participant deaths | 2 years and 5 years
Number of exacerbations as defined by a worsening of symptoms that warrant a change in medication. | 1 and 2 years
Number of hospital admissions | 1 and 2 years
Number of patients admitted to a nursing home | 2 and 5 years
Number of hospital bed days | 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, FRCP PhD, Principal Investigator — NIHR Respiratory Biomedical Research Unit Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Harefield hospital, Harefield, Middlesex, United Kingdom